CLINICAL TRIAL: NCT04501289
Title: Low Dose Magnesium Sulphate Versus Standard Pritchard Regimen In Management Of Severe Preeclampsia/Eclampsia: A Randomised Controlled Trial
Brief Title: Low Dose Magnesium Sulphate Versus Standard Pritchard Regimen In Management Of Severe Preeclampsia/Eclampsia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Adebayo Joshua Adeniyi (Other)
Responsible Party: Sponsor-Investigator, Adebayo Joshua Adeniyi, Doctor, Consultant, Department of Obstetrics and Gynaecology, Principal Investigator, Alex Ekwueme Federal University Teaching Hospital
Organization: Alex Ekwueme Federal University Teaching Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FETHA/REC/VOL1/2017/482
Record Dates: First submitted 2020-08-02; First posted 2020-08-06 (Actual); Last update posted 2020-08-06 (Actual); Status verified 2020-08

CONDITIONS: Preeclampsia/Eclampsia
Keywords: Preeclampsia; Eclampsia; Magnesium sulphate; Convulsion
MeSH Terms: conditions — Pre-Eclampsia; Eclampsia; Seizures | interventions — Magnesium Sulfate

STUDY DESIGN:
Intervention Model Description: The participants in the study will be randomized into two study groups in ratio 1:1. Participants in group 1 will receive 4g of 20% intravenous (I.V.) MgSO4, followed by 3g of 50% intramuscular (I.M.) MgSO4 in each buttock statim. Then, maintenance doses will be given as 2.5g of 50% MgSO4 I.M. 4 hourly for 24 hours, for patients with severe preeclampsia and for 24 hours post-delivery or post last seizure episode, for patients with eclampsia; while those in group 2 will receive loading dose as 4g of 20% MgSO4 I.V., followed by 5g of 50% MgSO4 I.M. in each buttock. Maintenance doses will be given as 5g of 50% MgSO4 I.M. 4 hourly in alternate buttock until 24 hours for participants with eclampsia and for 24 hours after delivery or after last fit, whichever occurs later, for those with eclampsia
Who Masked: Participant
Masking Description: Participants will be informed of the drug to be administered and the duration but were unaware of the dosage of the drug to be administered to them. However, the investigator knew the dosage each study cohort received
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low dose magnesium sulphate (Experimental): Experimental - participants in this arm will be pregnant women with severe preeclampsia/eclampsia who will receive low dose magnesium sulphate
  Interventions: Drug: Low dose magnesium sulphate
- Magnesium sulphate Pritchard regimen (Experimental): Experimental - participants in this arm will be pregnant women with severe preeclampsia/eclampsia who will receive Pritchard regimen of magnesium sulphate
  Interventions: Drug: Pritchard regimen

INTERVENTIONS:
Drug: Low dose magnesium sulphate — Participants in this arm will receive 4g of 20% intravenous (I.V.) MgSO4 (Magphate®) given over 10 minutes, followed by 3g of 50% intramuscular (I.M.) MgSO4 in each buttock statim. Then, maintenance doses will be given as 2.5g of 50% MgSO4 administered intramuscularly 4 hourly for 24 hours, for participants with severe preeclampsia and for 24 hours post delivery or post last seizure episode, whichever occurs last, for cohorts with eclampsia.
  Arms: Low dose magnesium sulphate
Drug: Pritchard regimen — Participants in this arm will receive loading dose as 4g of 20% MgSO4 I.V. over 10 minutes, followed by 5g of 50% MgSO4 I.M. in each buttock. Maintenance doses will be given as 5g of 50% MgSO4 I.M. 4 hourly in alternate buttock until 24 hours for patients with eclampsia and for 24 hours after delivery or after last fit, whichever occurs later, for cohorts with eclampsia.
  Arms: Magnesium sulphate Pritchard regimen

SUMMARY:
Background - Preeclampsia/eclampsia, a pregnancy specific multi-systemic disease, is associated with considerable maternal and perinatal morbidity and mortality. Prevention and/or treatment of convulsion with magnesium sulphate, among others, is life-saving. Despite different regimens that have been tried, the minimum effective dose of MgSO4 for the prevention of eclampsia in patients with preeclampsia and treatment of convulsion in those with eclampsia has not been determined.

Objectives - To compare the maternal and perinatal outcomes and maternal side effects in eclamptic and preeclamptic participants treated with low dose regimen of MgSO4 with those treated with the Pritchard regimen.

Materials and Methods - This will be a prospective, single blinded randomized controlled study of low dose versus Pritchard regimens of MgSO4. Participants will be randomly assigned to the either arm of the study. Efficacy and adverse effects of the drug on the mother and baby will be noted. Data will be collated, tabulated and then statistically analysed using the statistical package for social sciences (SPSS) Results - Conclusion will be drawn and recommendation made from the findings in the study.

DETAILED DESCRIPTION:
Introduction Preeclampsia complicates 5-7% of all pregnancies globally. However, hospital-based studies in Nigeria have reported rates ranging between 1.2% and 6.3%, while a study in Abakaliki recorded 0.99% for severe preeclampsia and 0.76% for eclampsia. Severe preeclampsia and eclampsia are associated with increased maternal and perinatal morbidity and mortality. The World Health Organization (WHO) estimates that about 63,000 maternal deaths occur annually from preeclampsia/eclampsia and associated complications, with 98% of these deaths occurring in developing countries. Perinatal adverse outcomes are usually due to prematurity associated with preterm delivery, as well as intrauterine fetal death from intrauterine growth restriction and placental abruption. Early recognition therefore, combined with prompt management, is often required for good maternal and perinatal outcome.

The definitive treatment for severe preeclampsia or eclampsia is delivery of the placenta. In affected women, positive maternal and perinatal outcomes depend on the woman having timely access to a treatment package which include effective inpatient monitoring, optimal timing of childbirth, presence of skilled attendant at birth and administration of antihypertensive as well as anticonvulsive therapy. Of all the anticonvulsants that have been tried in the management of preeclampsia and eclampsia, magnesium sulphate (MgSO4) has been established as the anticonvulsant of choice both for prevention of convulsions in severe preeclampsia and for prevention of recurrent convulsions in eclampsia. It has been shown to be superior to diazepam, phenytoin, and lytic cocktail (a mixture of chlorpromazine, promethazine and pethidine) in reducing the occurrence of eclamptic convulsion and the associated maternal morbidity and mortality. It also has beneficial effects on fetuses, reducing the risks of low Apgar scores in the 1st and 5th minutes, the risk of cerebral haemorrhage, as well as the need for intubation and admission into newborn intensive care units.

Magnesium sulphate belongs to the class of electrolytes anti-dysrrhythmic drugs. It is a sterile, non-pyrogenic concentrated solution of magnesium sulphate heptahydrate in water for injection. It is administered by the intravenous (IV) or intramuscular (IM) routes as an electrolyte replenisher or anticonvulsant. It has been adjudged to be the most effective, safe and low-cost anticonvulsant drug for pre-eclampsia and eclampsia. Though the mechanism of action is not completely understood, several hypotheses have been put forward to explain its beneficial effects in patients with preeclampsia and eclampsia. These include dilatation of cerebral blood vessels thereby reducing cerebral ischaemia, blockade of the N-methyl-D-aspartate receptors in the brain and also causing peripheral vasodilatation. However, despite its endorsement by the W.H.O. and its widespread availability, MgSO4 is still underused and incorrectly administered in many low resource settings. This has been discovered to be due to a number of provider factors and the complexity of treatment regimens being used.

The most commonly used MgSO4 regimens are those given intramuscularly and/or intravenously from the diagnosis of severe preeclampsia and eclampsia to 24 hours post delivery or post last seizure episode, whichever occurs later. Though these regimens have been found to be effective, they involve administering large doses of the drug. This usually leads to high cost of treatment to the affected patients as well as difficulties in monitoring such patients for drug toxicity (which include neurological deficit and cardiac arrest), especially in developing countries where manpower and facilities are limited. Therefore, several attempts have been made either to shorten the duration of administration or reduce the dosage of MgSO4 with the aim of achieving optimal efficacy, while reducing the side effects of the drug and the cost of management. These include those in which the loading dose and maintenance doses were reduced in quantities; those involving reduction of maintenance dose to 12 hours and those involving giving only the loading dose. No particular regimen has been generally adopted as the minimum effective dose, although several lower doses have proved to be effective. Because of their effectiveness which has been demonstrated over time, it has been suggested that lower doses of MgSO4 may suffice for prophylaxis for patients with severe preeclampsia as well as treatment for those with eclampsia, without jeopardising efficacy.

Though the reason for the success recorded with the low dose regimen used in Dhaka was attributed to the low body mass index of the population, several other studies in other places with varying dosages and different weight distribution have also recorded varying degrees of success. Therefore small body mass index (BMI) alone may not be enough to explain the whole phenomenon. Some authorities have also shown that there is no association between treatment failures and patients' BMI. or with serum magnesium levels. A systematic review in Nigeria in 2016 supported the fact that there were no studies that had demonstrated the lowest effective dose of MgSO4 to manage preeclampsia/eclampsia. Another systematic review also recommended further studies to identify the minimum effective dose of MgSO4 for the management of preeclampsia/eclampsia. Therefore, any regimen that will involve minimal cost and side effects; and at the same time be as effective as the current doses being administered, will go a long way in reducing the challenges of affordability of the drug and that of its side effects. It is against this background that this study is being carried out to compare the efficacy of a lower dose of MgSO4 in patients with severe pre-eclampsia and eclampsia to that of the Pritchard's regimen among our women population with a view to recommending it for use if the efficacy is found to be comparable.

Study background The study will be carried out at the Obstetric and Gynaecology division of Alex Ekwueme Federal University Teaching Hospital, Abakaliki, Ebonyi State, South-east, Nigeria. The department of Obstetrics and Gynaecology is one of the clinical departments in the hospital. There are 52 obstetric bed spaces including antenatal and postnatal wards. The department has five teams which are sub-divided into two units each. Each unit is manned by at least two consultants. Resident doctors are distributed to cover all the units. The department runs antenatal clinics managed by the consultants and resident doctors, assisted by midwives and other health workers. Antenatal clients are booked daily on every week day and are assigned consultants according to the units/teams running antenatal clinic each day. The average antenatal booking is about 4,200 clients per annum, while the total antenatal clinic attendance averages 21,000 per annum, with an average annual delivery rate of 3,100. The department has established protocols for management of specific cases which are in accordance with international best practices, and are displayed in the labour wards, antenatal ward and the accident and emergency unit of the hospital. These protocols serve as guides as patient care is still individualised.

For cases of severe preeclampsia and eclampsia, the departmental protocol is to stabilise the patient and deliver through the most expeditious route, though considerations may be given in certain cases of severe preeclampsia to allow for fetal growth for one or two weeks provided maternal and fetal clinical and laboratory parameters are stable. One of the steps taken during the period of stabilization is the administration of MgSO4 so as to avoid fits or its recurrence. The most commonly used MgSO4 regimen in the department is the Pritchard regimen in which MgSO4 is given as intravenous loading dose of 4g over 10 minutes, while 5g is administered intramuscularly in each buttock statim. Then 5g of MgSO4 is then administered intramuscularly every 4 hours until 24 hours after delivery or 24 hours after the last seizure episode, whichever occurs later, provided no sign of toxicity from the previous dose is noted. This is chosen because it involves less man-power for administration and monitoring of the patients.

Study population Participants to be included in this study will be women with severe preeclampsia and eclampsia that will be admitted and managed at the study facility who meet the inclusion criteria. Detailed history will be obtained and thorough examination will be carried out on all patients. Relevant investigations, which include blood group and Rhesus type, complete blood count, platelet count, liver function tests, kidney function tests, coagulation profile and urine analysis for proteinuria, will be carried out.

Sample size determination The minimum sample size will be determined using statistical formula for non-inferiority study design.

N= 2×[Z1-α/2+Z1-β]2 × P × (1-P) do N = number of patients per group Z = the standard normal deviate for a one or two sided study, usually set at 1.96.

d0 = clinically acceptable margin of equivalence which will be set at 0.05 P = proportion of patients in both arms who developed convulsion following administration of MgSO4 from a previous related study (0.2)50 α = type I error = ≤5% β = type II error =≤ 20% N = 2 × (1.96+0.845)2 × 0.2(1-0.2) 0.05 N = 2 × 7.868 × 0.2 × 0.8 0.05 N = 2.517768 0.05 N = 50.36 ≈ 50 This will represent the number of patients per group. Twenty percent of this minimum sample size will be added to correct for any attritions that may occur in the course of the study. The final sample size on each arm of the study will now be 60.

Participants' selection The participants will be randomized by means of a computer generated random numbers, by a statistician, using the software Research Randomizer®. Using this software, sixty numbers will be randomly generated from a pool of one hundred and twenty numbers (1-120) and these numbers will be assigned to group A (low dose) while the remaining sixty numbers will automatically be assigned to group B (Pritchard).

Group A: will receive 4g of 20% intravenous (I.V.) MgSO4 (Magphate®) given over 10 minutes, followed by 3g of 50% intramuscular (I.M.) MgSO4 in each buttock statim. Then, maintenance doses will be given as 2.5g of 50% MgSO4 administered intramuscularly 4 hourly for 24 hours, for those with severe preeclampsia and for 24 hours post delivery or post last seizure episode, whichever occurs last, for participantsts with eclampsia (low dose regimen).

Group B: will receive loading dose as 4g of 20% MgSO4 I.V. over 10 minutes, followed by 5g of 50% MgSO4 I.M. in each buttock. Maintenance doses will be given as 5g of 50% MgSO4 I.M. 4 hourly in alternate buttock until 24 hours for patients with eclampsia and for 24 hours after delivery or after last fit, whichever occurs later, for patients with eclampsia (Pritchard regimen).

These numbers (1-120) will be inscribed on brown envelopes and a piece of paper with the inscription 'low dose' or 'Pritchard' will be placed with the respective drug accordingly inside these envelopes and sealed. All the envelopes will be kept in a locker that will be made accessible to all the members of the research team. Participants will be made to know what the drug is meant to do for them during the counselling session and the possible side effects but will not know which arm of the study they belong (single blinding).

Participants, who meet the inclusion criteria, having signed the informed consent form, will be given sequential study numbers and the corresponding numbered opaque sealed envelope will then be allocated to the study cohorts.

Drug administration Participants allocated to the low dose arm, loading dose of magnesium sulphate will be administered starting with 4g of 20% MgSO4 I.M. over 10 minutes by the researcher/assistant, followed by 3g of 50% MgSO4 I.M. in each buttock statim. This will then be followed by administration of 2.5g of 50% MgSO4 I.M. 4 hourly in alternate buttock for 24 hours, for patients with severe preeclampsia and for 24 hours after delivery or last fit, whichever occurs later for patients with eclampsia. For those on the Prichard regimen, the loading dose will be given as 4g of 20% I.V. over 10 minutes, followed by 5g of 50% MgSO4 I.M. in each buttock. This will then be maintained by 5g of 50% I.M. MgSO4 4 hourly for 24 hours for patients with severe preeclampsia and for 24 hours after delivery or last convulsion, whichever occurs later, for cohorts with eclampsia. Participants' vital signs will be checked before MgSO4 administration. Toxicity will also be checked for as earlier outlined. If maintenance dose is found to be contraindicated in any of the patients based on her clinical status or presence of signs of toxicity, such participants will be excluded from the study. .

Monitoring Participants will be monitored clinically for signs of toxicity. This will be done by checking for deep tendon reflex which should be present, respiratory rate which should be not be less than 16 cycles per minute and hourly urine output which should be at least 30ml per hour. One gram of calcium gluconate will be provided for each patient on MgSO4 to be given in case of toxicity. For those who fit while on the low dose, 2g of 20% MgSO4 will be administered intravenously over 10 minutes while the patient is converted to the Pritchard regimen. Other causes of convulsion will also be sought for. If any of the participants on Pritchard regimen fits, she will be given 2g of 20% MgSO4 intravenously over 10 minutes while re-evaluating the woman for other possible causes of convulsion.

Statistical analysis Data will be collated, tabulated and then statistically analysed using the statistical package for social sciences (SPSS) (IBM) software (version 22, Chicago USA). Continuous variable will be presented as mean ± standard deviaton (SD), while categorical variables will be presented as numbers and percentages. Chi-square test will be used for comparison between groups of qualitative variables while normal z-test, risk ratio and confidence interval at 95% will be used for comparison between groups of quantitative variables. A difference with a p-value <0.05 will be considered statistically significant.

Ethical consideration Ethical clearance was obtained from the Research and Ethics committee of Alex Ekwueme Federal University Teaching Hospital, Abakaliki, Nigeria. A signed-written consent will be obtained from each participant before recruitment into the study. The participants will be made to understand that declining participation will have no consequences in her obtaining adequate care. The participants will be assured that their identity would be kept in confidence by the investigator.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with diagnosis of severe preeclampsia/eclampsia

Exclusion Criteria:

* Administration of MgSO4 before admission.
* Administration of diazepam or phenytoin before admission
* Maternal complications such as disseminated intravascular coagulation, cerebrovascular accident, renal disease, HELLP syndrome and aspiration pneumonitis.
* Multiple gestation
* Gestational ages below 28 weeks
* Postpartum eclampsia

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Pregnant women with gestational age of 28 weeks and above
Enrollment: 114 (Actual)
Dates: Start 2017-05-08 (Actual); Primary Completion 2017-12-27 (Actual); Study Completion 2018-01-22 (Actual)

PRIMARY OUTCOMES:
Convulsion | Within 24 hours of administration
  Occurrence of convulsion for participants with severe preeclampsia and recurrence of convulsion for cohorts with eclampsia

SECONDARY OUTCOMES:
Maternal side effects of MgSO4 | Within 24 hours of administration
  Deep tendon reflex
MgSO4 toxicity | Within 24 hours of administration
  Urine output less than 30ml/hr
Respiratory depression | Within 24 hours of administration
  Respiratory rate less than 12 cycles/min
Maternal complication 1 | Before delivery of baby
  Abruptio bplacentae
Maternal complication 2 | Within 24 hours of delivery
  Primary postpartum hemorrhage
Maternal complication 3 | Within 24 hours of delivery
  Mortality
Fetal outcome 1 | At delivery
  Apgar score
Fetal outcome 2 | At delivery
  Neonatal intensive care admission

CONTACTS AND LOCATIONS:
Overall Officials: Joshua A Adebayo, MB;BS; FWACS, Principal Investigator — Alex Ekwueme Federal University Teaching Hospital, Abakaliki
Locations (1):
- Alex Ekwueme Federal University Teaching Hospital, Abakaliki, Abakaliki LG, Nigeria

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data would be made available by the corresponding author on request
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 20 years